CLINICAL TRIAL: NCT03410082
Title: A Prospective Randomized Controlled Trial on the Patient's Satisfaction of Bispectral Index-guided Monitored Anesthesia Care
Brief Title: Patient's Satisfaction of Bispectral Index-guided Monitored Anesthesia Care
Acronym: BISMAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: extremely slow enrollment
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: snuhksm
Record Dates: First submitted 2017-07-26; First posted 2018-01-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Bispectral Index, Monitored Anesthesia Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The person who surveys the patient's satisfaction in the post anesthesia care unit does not know which group the patient was assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OAA/S (Active Comparator): The patients in the control group will receive MAC titrated according to observer's assessment of anesthesia/sedation(OAA/S) score.
  Interventions: Diagnostic Test: Titration under the guidance of OAA/S
- BIS (Active Comparator): The patients in the control group will receive MAC titrated according to bispectral index(BIS).
  Interventions: Device: Titration under the guidance of BIS

INTERVENTIONS:
Device: Titration under the guidance of BIS — The infusion rate of dexmedetomidine is increased by 0.1mcg/kg/h if BIS is greater than 80; The infusion rate is decreased by 0.1mcg/kg/h if BIS is less than 60.
  Arms: BIS
Diagnostic Test: Titration under the guidance of OAA/S — The infusion rate of dexmedetomidine is increased by 0.1mcg/kg/h if OAA/S is greater than 3; The infusion rate is decreased by 0.1mcg/kg/h if OAA/S is less than 3.
  Arms: OAA/S

SUMMARY:
The investigators will evaluate the effect of bispectral index-guided titration of sedation during ear surgery under monitored anesthesia care on participant's satisfaction with anesthesia, as well as side effects caused by the anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ear surgery with ASA physical status 1 or 2

Exclusion Criteria:

* Age under 19 years
* Pregnancy
* Cognitive disorder affecting daily activity
* Patients who cannot participate in the survey
* Allergy to the medication
* History of sedative abuse

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Iowa Satisfaction with Anesthesia Scale(ISAS) | within 30 minutes after the end of surgery (in the PACU)
  Patient's satisfaction with MAC

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Agree, South Korea

IPD SHARING:
Plan to Share IPD: No